CLINICAL TRIAL: NCT03275207
Title: a Randomized Controlled Trial of Dexmedetomidine on Chronic Postoperative Pain After Breast and Thoracic Surgery
Brief Title: Dexmedetomidine for Prevention of Chronic Postoperative Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Jian-jun Yang, director, department of anesthesiology, Zhongda Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 20170819
Record Dates: First submitted 2017-08-23; First posted 2017-09-07 (Actual); Last update posted 2017-12-05 (Actual); Status verified 2017-12

CONDITIONS: Chronic Postoperative Pain
Keywords: Chronic pain; CPSP; Dexmedetomidine; Surgery
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Sodium Chloride; Dexmedetomidine

STUDY DESIGN:
Intervention Model Description: paitents undergoing breast or thoracic surgery
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Placebo Comparator): an equal volume of saline
  Interventions: Drug: saline
- dexmedetomidine (Experimental): dexmedetomidine, 0.5ug/kg/h by intravenous infusion, intraoperative
  Interventions: Drug: dexmedetomidine

INTERVENTIONS:
Drug: saline — an equal volume of saline
  Arms: control group
Drug: dexmedetomidine — dexmedetomidine, 0.5ug/kg/h by intravenous infusion, intraoperative
  Arms: dexmedetomidine

SUMMARY:
Chronic postoperative pain (CPSP) is common symptom in patients after surgery, seriously affected the quality of life. Accumulating evidences have demonstrated dexmedetomidine can improve chronic pain. However, the prevention of dexmedetomidine on CPSP remain uncertain.

DETAILED DESCRIPTION:
Chronic postoperative pain (CPSP) is defined as pain persisting at least 3 months after surgery. It is most common in patients who undergoing breast or thoracic surgery. Dexmedetomidine, a adrenergic α2 agonists, can alleviate the postoperative pain 24 h after surgery. In our study, patients were randomly assigned to one of the two group to receive 0.5mg/kg/h infusion dexmedetomidine (Group D, n=57) or normal saline (Group C, n=57). The pain scales were evaluated day 1, day 2, day 3, month 3, month 6 after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have been 18 to 65 yr old, and been scheduled for breast or thoracic surgery.

Exclusion Criteria:

* Patients with limitations of self-expression or visual dysfunction or having emergency surgery, a severe psychiatric illness, or chronic pain problems in the chest area for longer than 2 months before the surgery,or patients who could not provide informed consent were excluded.
* Pregnant women and prisoners were also excluded.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2018-01-01 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-10-01 (Estimated)

PRIMARY OUTCOMES:
the pain intensity measure | 12 months
  Self reported pain intensity in rest and activity will be recorded at day 1 before sugery, month 3, month 6, month 12 after sugery. The intensity of pain was measured by numeric rating scale (0=no pain, 10=worst possible pain)

SECONDARY OUTCOMES:
anxiety | 12 months
  The anxiety will be self reported by patents at day 1 before surgery, month 3, month 6, month 12 after surgery.The anxiety will be scored by a Visual Analogue Scale of anxiety (0=no anxiety, 10=worst possible anxiety)
depression | 12 months
  The depression will be evaluated at day 1 before surgery, month 3, month 6, month 12 after sugery by a questionnaire
sleep disturbance | 12 months
  Sleep disturbance will be evaluated at day 1 before surgery, month 3, month 6, month 12 after sugery by questionnaires.

CONTACTS AND LOCATIONS:
Overall Officials: Yang Jian-jun, PhD, Principal Investigator — Zhongda Hospital
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No